CLINICAL TRIAL: NCT01788761
Title: The Effects of Probiotic Supplementation on Extremely Low Birthweight Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Health System (Network)
Collaborators: Rockford Memorial Hospital Development Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: pROBIOTICS11
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-04

CONDITIONS: Feeding Tolerance
Keywords: Probiotics; Feeding Tolerance; Extremely Low Birthweight Infants
MeSH Terms: interventions — Culture Techniques; Control Groups; Food, Formulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Supplemented Group (Experimental): 500,000,0000 cells of Lactobacillus GG (utilizing either Culturelle for Kids or Kids Culturelle preparation) and 500,000,000 cells of Bifidobacterium Infantis (utilizing Align capsule) diluted in 3 ml breastmilk/formula and administered enterally from first day of enteral feeds until term gestation/discharge/transfer/death (whichever occurs first) every day infant is receives enteral feedings
  Interventions: Dietary Supplement: Probiotic Supplemented Group
- Control Group (Sham Comparator): 3 ml enteral feeding of breastmilk/formula administered once daily in addition to regularly prescribed enteral feedings from day of first feeding until term gestation/discharge/transfer/death (which ever occurs first) and administered every day that infant receives enteral feedings
  Interventions: Dietary Supplement: Control Group

INTERVENTIONS:
Dietary Supplement: Probiotic Supplemented Group
  Other Names: Culture for Kids; Kids Culturelle; Align; Lactobacillus GG; Bifidobacter Infantis
  Arms: Probiotic Supplemented Group
Dietary Supplement: Control Group
  Other Names: Breastmilk; Formula
  Arms: Control Group

SUMMARY:
This is a research study that will look at the effects of giving two nutritional supplements on extremely low birth infants (infants weighing less than 1000 grams or weighing less than approximately 2 lbs 3 1/2 ounces at birth). The nutritional supplements that will be studied are Culturelle for Kids/Culturelle Kids and Align. They are nutritional supplements that each contain a different probiotic. In this study the investigators will mainly be looking at the effect that these supplements may have on how well babies tolerate their feedings and how long they require supplemental intravenous fluids for nutritional support. The investigators will also, however, look at many other factors such as rate of growth, rates of infection, survival rate and the length of time the infant needs to be in the hospital. The investigators will also look at its effect on conditions/complications of prematurity such as bronchopulmonary dysplasia and chronic lung disease (chronic diseases of the lung associated with prematurity), necrotizing enterocolitis and intestinal perforations (serious diseases of the infant's intestines), retinopathy of prematurity (eye disease associated with prematurity), intracranial hemorrhage (bleeding into the brain) and patent ductus arteriosus (a blood vessel connecting two main blood vessels coming out of the heart that does not close spontaneously (by itself).

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the effect of the administration of the nutritional supplements, Culturelle for Kids/Kids Culturelle in combination with Align, containing the Probiotics Lactobacillus GG and Bifidobacterium Infantis, on feeding tolerance (as determined by the number of days infant is without enteral feedings due to feeding intolerance, number of days infant requires supplemental hyperalimentation/intravenous fluids for nutritional support and number of days to achieve full enteral feedings) in high risk extremely low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight between 500-999 grams
* Apgar score greater than or equal to 3 at 5 minutes
* Infant free from any known major congenital anomalies or chromosomal/genetic anomalies
* Infant without any known cyanotic or complex congenital heart disease
* Infant NPO or on trophic enteral feedings than have been started less than 24 hours previously
* Infant without prior history of necrotizing enterocolitis or gastrointestinal perforation
* Infant without previous exposure to probiotics
* Infant that will be ready to start trophic feedings within the first 14 days of life
* Infant less than or equal to 14 days of age
* Infant born to HIV negative mother
* Written informed consent obtained from mother

Exclusion Criteria:

* Infant born to HIV positive mother
* Infant with history of prior probiotic exposure
* Infant greater than 14 days of age
* Infant on enteral feedings for greater than 24 hours
* Infant with major congenital anomaly/chromosomal or genetic anomaly
* Infant with cyanotic/complex congenital heart disease
* Infant with previous gastrointestinal perforation/necrotizing enterocolitis
* 5 minute Apgar score < 3

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2012-07; Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Feeding Tolerance | Evaluated on a daily basis until hospital discharge/transfer/death up until one year of age
  Feeding Tolerance as determined by the number of days infant is without enteral feedings due to feeding intolerance, number of days infant requires supplemental hyperalimentation/intravenous fluids for nutritional support and number of days to achieve full enteral feedings

SECONDARY OUTCOMES:
Necrotizing Enterocolitis (Bell's Stage 2 or greater) | Infants entire inpatient record assessed at/after time of hospital discharge/transfer/death up until 1 year of age
Culture proven sepsis without Necrotizing Enterocolitis | Infants entire inpatient record assessed at/after time of hospital discharge/transfer/death up until one year of age
Chronic Lung Disease | Infants entire inpatient record assessed at/after time of hospital discharge/transfer/death up until one year of age
Periventricular Leukomalacia | Infant's entire inpatient record assessed at/after time of hospital discharge/transfer/death up until one year of age
Mortality | Infant's entire inpatient record assessed at/after time of hospital discharge/transfer/death up until one year of age
Intraventricular Hemorrhage | Infants entire inpatient record assessed at/after time of hospital discharge/transfer/death up until one year of age
Daily weight gain in grams | Measured daily until time of hospital discharge/transfer/death up until one year of age
Discharge weight measured and expressed by percentile of growth for age | Assessed at the time of discharge/transfer/death up until one year of age
Length of Stay | Measured at time of discharge/transfer/death up until one year of age

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Schmidt, MS, APN, NNP, Principal Investigator — Mercy Health System
Locations (1):
- Rockford Memorial Hospital, Rockford, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfaleh K, Anabrees J, Bassler D. Probiotics reduce the risk of necrotizing enterocolitis in preterm infants: a meta-analysis. Neonatology. 2010;97(2):93-9. doi: 10.1159/000235684. Epub 2009 Aug 25. PMID 19707025
- [Background] Amerifit Inc. Culturelle Probiotics for Kids. Packaging information 2010
- [Background] Baldassarre ME, Laforgia N, Fanelli M, Laneve A, Grosso R, Lifschitz C. Lactobacillus GG improves recovery in infants with blood in the stools and presumptive allergic colitis compared with extensively hydrolyzed formula alone. J Pediatr. 2010 Mar;156(3):397-401. doi: 10.1016/j.jpeds.2009.09.012. Epub 2009 Nov 2. PMID 19880141
- [Background] Bin-Nun A, Bromiker R, Wilschanski M, Kaplan M, Rudensky B, Caplan M, Hammerman C. Oral probiotics prevent necrotizing enterocolitis in very low birth weight neonates. J Pediatr. 2005 Aug;147(2):192-6. doi: 10.1016/j.jpeds.2005.03.054. PMID 16126048
- [Background] Chou IC, Kuo HT, Chang JS, Wu SF, Chiu HY, Su BH, Lin HC. Lack of effects of oral probiotics on growth and neurodevelopmental outcomes in preterm very low birth weight infants. J Pediatr. 2010 Mar;156(3):393-6. doi: 10.1016/j.jpeds.2009.09.051. Epub 2009 Nov 14. PMID 19914635
- [Background] Dani C, Biadaioli R, Bertini G, Martelli E, Rubaltelli FF. Probiotics feeding in prevention of urinary tract infection, bacterial sepsis and necrotizing enterocolitis in preterm infants. A prospective double-blind study. Biol Neonate. 2002 Aug;82(2):103-8. doi: 10.1159/000063096. PMID 12169832
- [Background] Deshpande G, Rao S, Patole S, Bulsara M. Updated meta-analysis of probiotics for preventing necrotizing enterocolitis in preterm neonates. Pediatrics. 2010 May;125(5):921-30. doi: 10.1542/peds.2009-1301. Epub 2010 Apr 19. PMID 20403939
- [Background] Guenther K, Straube E, Pfister W, Guenther A, Huebler A. Sever sepsis after probiotic treatment with Escherichia coli NISSLE 1917. Pediatr Infect Dis J. 2010 Feb;29(2):188-9. doi: 10.1097/INF.0b013e3181c36eb9. No abstract available. PMID 20118747
- [Background] Indrio F, Riezzo G, Raimondi F, Bisceglia M, Cavallo L, Francavilla R. Effects of probiotic and prebiotic on gastrointestinal motility in newborns. J Physiol Pharmacol. 2009 Dec;60 Suppl 6:27-31. PMID 20224148
- [Background] Hojsak I, Abdovic S, Szajewska H, Milosevic M, Krznaric Z, Kolacek S. Lactobacillus GG in the prevention of nosocomial gastrointestinal and respiratory tract infections. Pediatrics. 2010 May;125(5):e1171-7. doi: 10.1542/peds.2009-2568. Epub 2010 Apr 19. PMID 20403940
- [Background] Kuitunen M, Kukkonen K, Savilahti E. Pro- and prebiotic supplementation induces a transient reduction in hemoglobin concentration in infants. J Pediatr Gastroenterol Nutr. 2009 Nov;49(5):626-30. doi: 10.1097/MPG.0b013e31819de849. PMID 19644396
- [Background] Ladd N, Ngo T. The use of probiotics in the prevention of necrotizing enterocolitis in preterm infants. Proc (Bayl Univ Med Cent). 2009 Jul;22(3):287-91. doi: 10.1080/08998280.2009.11928535. No abstract available. PMID 21240300
- [Background] Lin HC, Su BH, Chen AC, Lin TW, Tsai CH, Yeh TF, Oh W. Oral probiotics reduce the incidence and severity of necrotizing enterocolitis in very low birth weight infants. Pediatrics. 2005 Jan;115(1):1-4. doi: 10.1542/peds.2004-1463. PMID 15629973
- [Background] Lin HC, Hsu CH, Chen HL, Chung MY, Hsu JF, Lien RI, Tsao LY, Chen CH, Su BH. Oral probiotics prevent necrotizing enterocolitis in very low birth weight preterm infants: a multicenter, randomized, controlled trial. Pediatrics. 2008 Oct;122(4):693-700. doi: 10.1542/peds.2007-3007. PMID 18829790
- [Background] Luoto R, Isolauri E, Lehtonen L. Safety of Lactobacillus GG probiotic in infants with very low birth weight: twelve years of experience. Clin Infect Dis. 2010 May 1;50(9):1327-8. doi: 10.1086/651694. No abstract available. PMID 20367236
- [Background] Ohishi A, Takahashi S, Ito Y, Ohishi Y, Tsukamoto K, Nanba Y, Ito N, Kakiuchi S, Saitoh A, Morotomi M, Nakamura T. Bifidobacterium septicemia associated with postoperative probiotic therapy in a neonate with omphalocele. J Pediatr. 2010 Apr;156(4):679-81. doi: 10.1016/j.jpeds.2009.11.041. PMID 20303445
- [Background] Rinne M, Kalliomaki M, Arvilommi H, Salminen S, Isolauri E. Effect of probiotics and breastfeeding on the bifidobacterium and lactobacillus/enterococcus microbiota and humoral immune responses. J Pediatr. 2005 Aug;147(2):186-91. doi: 10.1016/j.jpeds.2005.03.053. PMID 16126047
- [Background] Rouge C, Piloquet H, Butel MJ, Berger B, Rochat F, Ferraris L, Des Robert C, Legrand A, de la Cochetiere MF, N'Guyen JM, Vodovar M, Voyer M, Darmaun D, Roze JC. Oral supplementation with probiotics in very-low-birth-weight preterm infants: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2009 Jun;89(6):1828-35. doi: 10.3945/ajcn.2008.26919. Epub 2009 Apr 15. PMID 19369375
- [Background] Salminen S, Collado MC, Isolauri E, Gueimonde M. Microbial-host interactions: selecting the right probiotics and prebiotics for infants. Nestle Nutr Workshop Ser Pediatr Program. 2009;64:201-13; discussion 213-7, 251-7. doi: 10.1159/000235792. Epub 2009 Aug 19. PMID 19710524
- [Background] Samanta M, Sarkar M, Ghosh P, Ghosh Jk, Sinha Mk, Chatterjee S. Prophylactic probiotics for prevention of necrotizing enterocolitis in very low birth weight newborns. J Trop Pediatr. 2009 Apr;55(2):128-31. doi: 10.1093/tropej/fmn091. Epub 2008 Oct 8. PMID 18842610
- [Background] Scalabrin DM, Johnston WH, Hoffman DR, P'Pool VL, Harris CL, Mitmesser SH. Growth and tolerance of healthy term infants receiving hydrolyzed infant formulas supplemented with Lactobacillus rhamnosus GG: randomized, double-blind, controlled trial. Clin Pediatr (Phila). 2009 Sep;48(7):734-44. doi: 10.1177/0009922809332682. Epub 2009 Mar 4. PMID 19264721
- [Background] Schanler RJ. Probiotics and necrotising enterocolitis in premature infants. Arch Dis Child Fetal Neonatal Ed. 2006 Nov;91(6):F395-7. doi: 10.1136/adc.2005.092742. No abstract available. PMID 17056837
- [Background] Soll RF. Probiotics: are we ready for routine use? Pediatrics. 2010 May;125(5):1071-2. doi: 10.1542/peds.2010-0643. Epub 2010 Apr 26. No abstract available. PMID 20421256
- [Background] Tarnow-Mordi WO, Wilkinson D, Trivedi A, Brok J. Probiotics reduce all-cause mortality and necrotizing enterocolitis: it is time to change practice. Pediatrics. 2010 May;125(5):1068-70. doi: 10.1542/peds.2009-2151. Epub 2010 Apr 19. No abstract available. PMID 20403934
- [Background] Anderson, T., Lord, A., Shotkoski, N. and O'Keefe, C. The use of probioitics for the prevention of necrotizing enterocolitis in the premature infant. Infant, Child and Adolescent Nutrition 2009; October: 246-249.